CLINICAL TRIAL: NCT06820398
Title: Effects of Functional Exercise Program With Strength Load and Resistance in Gross Motor Function, Quality of Life and Participation in Children and Adolescents With Cerebral Palsy Levels III-IV GMFCS
Brief Title: Effects of Functional Exercise Program With Strength Load and Resistance in Children and Adolescents With Cerebral Palsy
Acronym: FESCA_CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, M Luz Sanchez, Associate Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3498583
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
Keywords: Functional Exercise; Strength; Resistance; Children; Adolescents
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional exercise with progressive strength and resistance load (Experimental): This group will perform functionalexercises with progressive strengthand resistance load, adjusted basedon heart rate.
  Interventions: Other: Functional exercise with progressive strength and resistance load
- Functional exercises without any load (Active Comparator): This group will perform functionalexercises without strength orresistance load.
  Interventions: Other: Functional exercises without any load

INTERVENTIONS:
Other: Functional exercise with progressive strength and resistance load — This group will perform functional exercises with progressive strength and resistance load, adjusted based on heart rate.
  Arms: Functional exercise with progressive strength and resistance load
Other: Functional exercises without any load — This group will perform functional exercises, without strength or resistance load
  Arms: Functional exercises without any load

SUMMARY:
This research project aims to evaluate the benefits of a functional exercise program with strength and resistance load in adolescents with cerebral palsy (CP), specifically classifiedat levels III and IV of the Gross Motor Function Classification System (GMFCS) scale. Participants will be included into control or intervention group in this randomized controlled trial. Changes in functional percentile, quality of life, and participation in daily environments will be analyzed based on scores obtained with validated assesment scales.

The study will be conducted at the Children's Neurorehabilitation Unit of Hospitalarias Foundation in Valencia, with an 18-week intervention plus a 6-month follow-up. This project seeks to provide evidence on rehabilitation strategies that promote autonomy and social inclusion for this population.

DETAILED DESCRIPTION:
This research project is a randomized controlled trial designed to analyze the effects of a functional exercise program with strength and resistance load in adolescents with CP specifically classified at levels III and IV of the GMFCS scale. The study will include around 40 participants aged 10 to 18 years, randomly assigned to either an intervention group or a control group. The intervention group will perform functional exercises with progressive strength and resistance load, adjusted based on heart rate. The control group will perform the same functional exercises but without any load.

The protocol includes 36 sessions over 18 weeks, with evaluations at three key time points: before the intervention, at the end of the protocol, and six months post-intervention. The primary outcomes include functional percentile within the GMFCS, quality of life asperceived by patients and caregivers, and participation in daily environments.

The study will adhere to CONSORT guidelines and the Declaration of Helsinki and has been reviewed by an ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10 to 18 years.
* Diagnosis of spastic cerebral palsy (CP).
* Classification at levels III or IV of the GMFCS scale.

Exclusion Criteria:

* Multilevel surgery with osteotomy within the last 12 months.
* Microtenotomies or percutaneous needle lengthening (APAI) within the last 9months.
* Botulinum toxin injections within the last 3 months.
* Participation in specific strength training protocols.
* Lack of cognitive ability to perform the intervention protocol activities.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Percentile Based on Gross Motor Function Classification System (GMFCS) | Baseline (pre-intervention) and immediately post-intervention (at 18 weeks).
  This variable represents the functional percentile calculated using the Gross Motor Function Classification System (GMFCS) and related measures. It incorporates: 1)GMFCS: A five-level system classifying gross motor movement capacity; 2) GrossMotor Function Measure (GMFM-66 and GMFM-88): Tools for evaluating grossmotor function across multiple dimensions; and 3) GMAE-2 Software: Generatesfunctional percentiles based on GMFM data. Values range from 0 to 100, where 0 represents the lowest functional percentile and 100 the highest.

SECONDARY OUTCOMES:
Quality of Life Assessed with CP-QOL Questionnaire | Baseline (pre-intervention) and immediately post-intervention (at 18 weeks).
  This variable evaluates the quality of life of caregivers and adolescents using theCerebral Palsy Quality of Life Questionnaire (CP-QOL). The questionnaireassesses multiple domains of well-being and quality of life related to cerebral palsy.Values depend on the raw or normalized scores, which may vary depending on thescoring method. If normalized, scores range from 0 (lowest quality of life) to 100(highest quality of life).
Participation in Daily Environments Assessed with PEM-CY | Baseline(pre-intervention) and immediately post-intervention (at 18 weeks).
  This variable measures the participation of children and adolescents aged 5-18years in daily environments using the Participation and Environment Measure forChildren and Youth (PEM-CY). The PEM-CY evaluates both the frequency ofparticipation in various activities and the impact of environmental factors. Valuesare reported on scales specific to PEM-CY domains, where higher scores indicategreater participation and/or better environmental support.
Baseline Heart Rate | Baseline (pre-intervention) and immediately post-intervention (at 18 weeks).
  This variable represents the baseline heart rate, measured in beats per minute(bpm). It is recorded under resting conditions prior to any intervention or physicalactivity. Values range from 40 to 120 bpm, where lower values are associated withgreater tolerance to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: M.Luz Sánchez-Sánchez, PhD, Study Director — University of Valencia; Juan Francisco Lison Párraga, PhD, Study Director — Cardenal Herrera University; María Dolores Arguisuelas Martínez, PhD, Study Director — Cardenal Herrera University
Locations (1):
- Faculty of Physiotherapy. University of Valencia, Valencia, Spain